CLINICAL TRIAL: NCT04354376
Title: Replication of the TRANSCEND Antihypertensive Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-TRANSCEND
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Sodium Potassium Chloride Symporter Inhibitors; Thiazides; Dihydropyridines; Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Loop diuretics, thiazides, dihydropyridines: Reference group
  Interventions: Drug: Loop diuretics, thiazides, dihydropyridines
- Telmisartan: Exposure group
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Loop diuretics, thiazides, dihydropyridines — Loop diuretics, thiazides, or dihydropyridines dispensing claim is used as the reference
  Groups: Loop diuretics, thiazides, dihydropyridines
Drug: Telmisartan — Telmisartan dispensing claim is used as the exposure
  Groups: Telmisartan

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Please see: https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

The patients will be required to have continuous enrollment during baseline period of 180 days before initiation of telmisartan or a comparator drug (cohort entry).

Eligible cohort entry dates: Market availability of telmistartan in the U.S. started on November 10, 1998, however, the Marketscan and Optum data are available at BWH only from Jan 1, 2003 and Jan 1, 2004, respectively.

For Marketscan: Jan 1, 2003 -Dec 2017 (end of data availability). For Optum: Jan 1, 2004-June 30, 2019 (end of data availability).

Inclusion Criteria:

* Individuals 55 years of age with 1 of the following:

  * 1. Coronary artery disease

    * 1a. Previous myocardial infraction ( > 2 days post uncomplicated MI)
    * 1b. Stable angina or unstable angina > 30 days before informed consent and with documented evidence of multivessel coronary artery disease
    * 1c. Multi-vessel PTCA >30 days before informed consent
    * 1d. Multi-vessel CABG surgery > 4 years before informed consent, or with recurrent angina following surgery
  * 2. Peripheral artery disease

    * 2a. Previous limb bypass surgery or Previous limb bypass surgery or angioplasty
    * 2b. Previous limb or foot amputation
    * 2c. Intermittent claudication, with ankle:arm BP ratio =< 0.80 on at least 1 side
    * 2d. Significant peripheral artery stenosis ( > 50%) documented by angiography or non-invasive testing
  * 3. Cerebrovascular disease

    * 3a. Previous stroke
    * 3b. Transient ischemic attacks >7 days and <1 year before informed consent
  * 4. Diabetus mellitus

    * 4a. Diabetes mellitus High-risk diabetics with evidence of endorgan damage

Exclusion Criteria:

* 1. Medication use

  * 1a. Inability to discontinue ACE inhibitors or ARB
  * 1b. Known hypersensitivity or intolerance to ACE inhibitors or ARB (patient intolerant of ACE inhibitor can be enrolled in TRANSCEND)
* 2. Cardiovascular disease (HF)

  * 2a. Symptomatic congestive heart failure
  * 2b. Hemodynamically significant primary valvular or outflow tract obstruction
  * 2c. Constrictive pericarditis
  * 2d. Complex congenital heart disease
  * 2e. Syncopal episodes of unknown etiology <3 months before informed consent
  * 2f. Planned cardiac surgery or PTCA <3 months of informed consent
  * 2g. Uncontrolled hypertension on treatment (eg, BP >160/100 mm Hg)
  * 2f. Heart transplant recipient
  * 2g. Stroke due to subarachnoid hemorrhage
* 3. Other conditions

  * 3a. Significant renal artery disease
  * 3b. Hepatic dysfunction
  * 3c. Uncorrected volume or sodium depletion
  * 3d. Primary hyperaldosteronism
  * 3e. Hereditary fructose intolerance
  * 3f. Other major noncardiac illness expected to reduce life expectancy or interfere with study participation
  * 3g. Simultaneously taking another experimental drug
  * 3h. Significant disability precluding regular follow-up visits
  * 3I. Unable or unwilling to provide written informed consent

Min Age: 55 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, propensity score-matched, retrospective cohort study design comparing telmisartan to other antihypertensives, including loop diuretics, thiazides, and dihydropyridines. Although the trial compared telmisartan with placebo added to usual care, the investigators selected an active comparator for this study because non-user comparator groups are known to often lead to confounding by indication and biased treatment effect estimates. This group of other antihypertensives were selected as the primary comparator because intolerance to ACEi was a primary inclusion criteria for the trial. Therefore, patients in both arms were on a mix of non-ACEi and non-ARB antihypertensives as background therapy.
Sampling Method: Probability Sample
Enrollment: 40048 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Relative hazard of composite outcome of Congestive Heart Failure, Stroke, MI, and Mortality | Through study completion (a median of ***118-123**** days)
  Relative hazard of composite outcome of Congestive Heart Failure, Stroke, MI, and Mortality - Please refer to uploaded protocol for full definition due to size limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham And Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT04354376/Prot_SAP_001.pdf